CLINICAL TRIAL: NCT03719521
Title: Community Based Interventions to Improve HIV Outcomes in Youth: a Cluster Randomised Trial in Zimbabwe (CHIEDZA)
Brief Title: Community Based Interventions to Improve HIV Outcomes in Youth: a Cluster Randomised Trial in Zimbabwe
Acronym: CHIEDZA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Biomedical Research and Training Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16124
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: HIV Infection
Keywords: Adolescents; Youth; Sexual and reproductive health; Africa; community-based
MeSH Terms: conditions — HIV Infections; Coitus

STUDY DESIGN:
Intervention Model Description: Community Based Interventions to improve HIV outcomes in youth: a cluster randomised trial
Who Masked: Outcomes Assessor
Masking Description: Staff conducting the outcome survey will be masked to the arm allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Community-based provision of an integrated package of services over a 24 month period.
  For all those aged 16-24 years residing in the intervention clusters: HIV testing, Sexual and reproductive health services (condoms, menstrual hygiene management, contraception, syndromic sexually transmitted infection (STI) treatment, referral for voluntary medical male circumcision, cervical screening), General health information and counselling. For those who are aged 16-24 years and test HIV-positive (or known HIV positive) within the intervention clusters: ART initiation and community-based treatment, adherence support.
  Interventions: Other: Community-based package of integrated HIV, SRH and general health services
- Control Arm (Active Comparator): Routine existing services
  Interventions: Other: Community-based package of integrated HIV, SRH and general health services

INTERVENTIONS:
Other: Community-based package of integrated HIV, SRH and general health services — HIV Testing and Counselling, SRH and HIV prevention Services and General Health Counselling for all 16-24 year olds and ART initiation and ongoing treatment and adherence support for those who test HIV positive
  Other Names: Cluster-randomized trial

SUMMARY:
A cluster randomised trial to determine the impact of an integrated community-based package of HIV services incorporating HIV testing, linkage to care and ongoing adherence support, combined with sexual and reproductive health (SRH) services and general health counselling for 16 to 24 year olds on population level HIV viral load in a high HIV prevalence setting.

DETAILED DESCRIPTION:
Young people fare disproportionately poorly across the HIV care continuum compared to other age-groups; the prevalence of undiagnosed HIV is substantially higher, and coverage of and adherence to antiretroviral therapy is lower, resulting overall in worse virological outcomes.

Aim: The aim is to determine the impact of an integrated community-based package of HIV services incorporating HIV testing, linkage to care and ongoing adherence support, combined with sexual and reproductive health services and general health counselling for 16 to 24 year olds on population level HIV viral load in a high HIV prevalence setting.

Design: This is a two-arm cluster-randomised trial in 24 clusters randomised 1:1 to standard of care or to the intervention package.

Intervention: Community-based package of services that includes: HIV testing and counselling, delivery of antiretroviral therapy, adherence support groups, mobile health, condoms, menstrual hygiene management, contraception and treatment of sexually transmitted infections, referral for voluntary medical male circumcision and cervical screening, risk reduction counselling and general health information and counselling. The intervention will be implemented over a two and half year period. The intervention will be implemented in 12 clusters, each with a population of approximately 2500-4000 16-24 year olds.

Study Outcomes: The study outcomes will be determined at a population level through a community cross-sectional survey among 18 to 24 year olds two years following the implementation of the intervention. The primary outcome is the proportion with HIV with a viral load <1000 copies/ml. The secondary outcomes will reflect each step of the HIV care cascade: proportion with HIV who know their HIV status, proportion of those who know their HIV-positive status who are currently taking antiretroviral therapy, proportion of those taking antiretroviral therapy who are virally suppressed. Sexual and reproductive health knowledge, risks and behaviour will also be assessed.

Study population: The end-line survey will recruit 700 18-24 year olds per cluster (total 16 800).

Study sites: The study will be conducted in 3 provinces in Zimbabwe: Harare, Bulawayo and Mashonaland East.

Study Duration: The planned duration of the entire study will be 4 years

ELIGIBILITY:
Inclusion Criteria:

* Reside within cluster boundaries
* Aged 16 to 24 years

Exclusion Criteria:

* Reside outside the cluster boundaries
* Aged below 16 years
* Aged above 24 years

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36991 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Viral suppression among HIV-positive individuals | Measured after the 30 months of intervention.
  % of those with HIV with an HIV viral load <1000 copies /ml

SECONDARY OUTCOMES:
Knowledge of HIV-positive status | After 30 months of intervention
  % with an HIV-positive test who know they are HIV-positive
Coverage of antiretroviral therapy (ART) among those who their positive HIV status | After 30 months of the intervention
  % of those who know their positive HIV status who are currently taking ART
Viral suppression among those who report taking ART | After 30 months of the intervention
  % of those taking ART who have an HIV viral load <1000 copies /ml

CONTACTS AND LOCATIONS:
Overall Officials: Rashida Ferrand, PhD, Principal Investigator — LondonSchool Of Hygiene and Tropical Medicine
Locations (3):
- Zimbabwe (3):
  - Mashonaland East Province, Marondera, Mashonaland East Province
  - Bulawayo Province, Bulawayo
  - Harare Province, Harare

IPD SHARING:
Plan to Share IPD: Yes
Data will be placed in the London School of Hygiene and Tropical Medicine (LSHTM) research data repository. This repository will enable direct download of records with codebooks to enable replication of the data analyses. Data will be anonymised prior to release for data sharing. In addition, annotated questionnaires and STATA do-files used for data cleaning and analysis will be available. All databases will be password-protected and accessible to authorised personnel only. The LSHTM open access repository will also enable access to repository contents through a searchable index.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol and consent forms will be shared as soon as approved by ethical review boards. The clinical study report will be available on completion of the end line survey and the analytic code will be available 12 months after completion of the study
Access Criteria: Where individual data are concerned, the informed consent procedure will clarify the possibility of use of anonymised data by other researchers. Data users will be required to acknowledge the source of data and to ensure that the regulatory requirements of the Medical Research Council of Zimbabwe and other ethical bodies reviewing the projects are met.
URL: http://datacompass.lshtm.ac.uk/

REFERENCES:
- [Derived] Simms V, Dauya E, Dziva Chikwari C, Bandason T, Kranzer K, Tembo M, Mavodza C, Doyle AM, Larsson L, Mugurungi O, Apollo T, Hayes RJ, Ferrand RA; CHIEDZA trial team. Uptake of community-based integrated HIV and sexual and reproductive health services for young people in Zimbabwe: the CHIEDZA study. BMC Health Serv Res. 2025 Nov 10;25(1):1459. doi: 10.1186/s12913-025-13635-3. PMID 41214672
- [Derived] Ferrand RA, Dauya E, Chikwari CD, Bandason T, Bernays S, Mackworth-Young C, Doyle AM, Grundy C, Indravudh P, Terris-Presholt F, Mavodza CV, Mugurungi O, Apollo T, Ncube G, Larsson L, McCarthy O, Simms V, Tembo M, Kranzer K, Hayes RJ. Integrated community-based HIV and sexual and reproductive health services for youth: a cluster-randomized trial. Nat Med. 2025 Sep;31(9):3081-3088. doi: 10.1038/s41591-025-03762-z. Epub 2025 Jun 24. PMID 40555749
- [Derived] Kelly SH, Azizi S, Chikwari CD, Tembo M, Bandason T, Dauya E, Mavodza CV, Apollo T, Mugurungi O, Ferrand RA, Simms V. Awareness, access to and uptake of HIV prevention interventions among youth in Zimbabwe: a population-based survey. BMC Infect Dis. 2025 May 16;25(1):709. doi: 10.1186/s12879-025-11076-1. PMID 40380099
- [Derived] Dziva Chikwari C, Dauya E, Simms V, Kranzer K, Bandason T, Machiha A, Mugurungi O, Musiyandaka P, Mwaturura T, Tshuma N, Bernays S, Mavodza C, Tembo M, Martin K, Mackworth-Young CRS, Busza J, Francis SC, Hayes RJ, Ferrand RA. Effect of a community-based intervention for sexually transmitted infections on population-level prevalence among youth in Zimbabwe (STICH): a cluster-randomised trial. Lancet Glob Health. 2025 Jan;13(1):e134-e145. doi: 10.1016/S2214-109X(24)00373-5. Epub 2024 Nov 14. PMID 39551057
- [Derived] Hlahla K, Azizi SC, Simms V, Dziva Chikwari C, Dauya E, Bandason T, Tembo M, Mavodza C, Kranzer K, Ferrand R. Prevalence of substance and hazardous alcohol use and their association with risky sexual behaviour among youth: findings from a population-based survey in Zimbabwe. BMJ Open. 2024 Jun 16;14(6):e080993. doi: 10.1136/bmjopen-2023-080993. PMID 38885985
- [Derived] Martin K, Dauya E, Simms V, Bandason T, Azizi S, Machiha A, Shamu T, Musiyandaka P, Mwaturura T, Francis SC, Mackworth-Young CRS, Busza J, Mavodza C, Tembo M, Hayes RJ, Kranzer K, Ferrand RA, Dziva Chikwari C. Risk factors for curable sexually transmitted infections among youth: findings from the STICH population survey in Zimbabwe. Sex Transm Infect. 2024 Nov 18;100(8):484-491. doi: 10.1136/sextrans-2024-056146. PMID 38871454
- [Derived] Dziva Chikwari C, Kranzer K, Simms V, Patel A, Tembo M, Mugurungi O, Sibanda E, Mufare O, Ndlovu L, Muzangwa J, Vundla R, Chibaya A, Hayes R, Mackworth-Young C, Bernays S, Mavodza C, Hove F, Bandason T, Dauya E, Ferrand RA. Differentiated care for youth in Zimbabwe: Outcomes across the HIV care cascade. PLOS Glob Public Health. 2024 Feb 21;4(2):e0002553. doi: 10.1371/journal.pgph.0002553. eCollection 2024. PMID 38381752
- [Derived] Dziva Chikwari C, Dauya E, Bandason T, Tembo M, Mavodza C, Simms V, Mackworth-Young CR, Apollo T, Grundy C, Weiss H, Kranzer K, Mavimba T, Indravudh P, Doyle A, Mugurungi O, Machiha A, Bernays S, Busza J, Madzima B, Terris-Prestholt F, McCarthy O, Hayes R, Francis S, Ferrand RA. The impact of community-based integrated HIV and sexual and reproductive health services for youth on population-level HIV viral load and sexually transmitted infections in Zimbabwe: protocol for the CHIEDZA cluster-randomised trial. Wellcome Open Res. 2023 Nov 7;7:54. doi: 10.12688/wellcomeopenres.17530.2. eCollection 2022. PMID 38162283
- [Derived] Mavodza CV, Bernays S, Mackworth-Young CRS, Nyamwanza R, Nzombe P, Dauya E, Chikwari CD, Tembo M, Apollo T, Mugurungi O, Madzima B, Nguwo D, Ferrand RA, Busza J. Fidelity, Feasibility and Adaptation of a Family Planning Intervention for Young Women in Zimbabwe: Provider Perspectives and Experiences. Glob Implement Res Appl. 2023;3(2):182-194. doi: 10.1007/s43477-023-00075-6. Epub 2023 Mar 24. PMID 37293631
- [Derived] Tembo M, Weiss HA, Larsson LS, Bandason T, Redzo N, Dauya E, Nzanza T, Ishumael P, Gweshe N, Ndlovu P, Dziva Chikwari C, Mavodza CV, Renju J, Francis SC, Ferrand R, Mackworth-Young CRS. A mixed-methods study measuring the effectiveness of a menstrual health intervention on menstrual health knowledge, perceptions and practices among young women in Zimbabwe. BMJ Open. 2023 Mar 9;13(3):e067897. doi: 10.1136/bmjopen-2022-067897. PMID 36894201
- [Derived] Mavodza CV, Bernays S, Mackworth-Young CRS, Nyamwanza R, Nzombe P, Dauya E, Dziva Chikwari C, Tembo M, Apollo T, Mugurungi O, Madzima B, Kranzer K, Abbas Ferrand R, Busza J. Interrupted Access to and Use of Family Planning Among Youth in a Community-Based Service in Zimbabwe During the First Year of the COVID-19 Pandemic. Stud Fam Plann. 2022 Sep;53(3):393-415. doi: 10.1111/sifp.12203. Epub 2022 Jun 22. PMID 35731634
- [Derived] Tembo M, Renju J, Weiss HA, Dauya E, Gweshe N, Ndlovu P, Nzombe P, Chikwari CD, Mavodza CV, Mackworth-Young CRS, A Ferrand R, Francis SC. Integration of a menstrual health intervention in a community-based sexual and reproductive health service for young people in Zimbabwe: a qualitative acceptability study. BMC Health Serv Res. 2022 Mar 30;22(1):421. doi: 10.1186/s12913-022-07818-5. PMID 35354445
- [Derived] Martin K, Dziva Chikwari C, Mackworth-Young CRS, Chisenga M, Bandason T, Dauya E, Olaru ID, Francis SC, Mavodza C, Nzombe P, Nyamwanza R, Hove F, Tshuma M, Machiha A, Kranzer K, Ferrand RA. "It was difficult to offer same day results": evaluation of community-based point-of-care testing for sexually transmitted infections among youth using the GeneXpert platform in Zimbabwe. BMC Health Serv Res. 2022 Feb 10;22(1):171. doi: 10.1186/s12913-022-07557-7. PMID 35144602
- [Derived] Mavodza CV, Mackworth-Young CRS, Bandason T, Dauya E, Chikwari CD, Tembo M, Apollo T, Ncube G, Kranzer K, Ferrand RA, Bernays S. When healthcare providers are supportive, 'I'd rather not test alone': Exploring uptake and acceptability of HIV self-testing for youth in Zimbabwe - A mixed method study. J Int AIDS Soc. 2021 Sep;24(9):e25815. doi: 10.1002/jia2.25815. PMID 34569710
- [Derived] Tembo M, Renju J, Weiss HA, Dauya E, Bandason T, Dziva-Chikwari C, Redzo N, Mavodza C, Losi T, Ferrand R, Francis SC. Menstrual product choice and uptake among young women in Zimbabwe: a pilot study. Pilot Feasibility Stud. 2020 Nov 23;6(1):182. doi: 10.1186/s40814-020-00728-5. PMID 33292659